CLINICAL TRIAL: NCT07185672
Title: PReCedeNT Trial: Phase III Randomised Controlled Open Label Trial of Lutetium 177 PRRT Plus Chemotherapy Versus PRRT Aalone in FDG Avid Well Differentiated Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: PRRT Versus PRRT Plus Chemotherapy in GEP NET (PReCedeNT Trial)
Acronym: PReCedeNT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Ameya Puranik, Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMCIEC3258
Record Dates: First submitted 2025-08-25; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Neoplasia's (NENs); Neuroendocrine Tumor GEP Grade 1-3; Neuroendocrine Gastroenteropancreatic Tumour
Keywords: Peptide Receptor Radionuclide Therapy; Lu-177 DOTATATE; PRRT; Neuroendocrine tumor; Capecitabine-Temozolamide
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Phase 3 Open label Parallel Group Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peptide Receptor Radionuclide Therapy with Lu177 DOTATATE (Active Comparator): Patient in this arm will be treated only with 4 cycles of PRRT
  Interventions: Radiation: Peptide Receptor Radionuclide Therapy with Lu177 DOTATATE
- PRRT with Lu-177 DOTATATE PLUS Capecitabine-Temozolamide (Experimental): Patient in this arm will be treated with combination of PRRT and Chemotherapy
  Interventions: Radiation: Peptide Receptor Radionuclide Therapy with Lu177 DOTATATE; Drug: Capecitabine plus temozolamide

INTERVENTIONS:
Radiation: Peptide Receptor Radionuclide Therapy with Lu177 DOTATATE — Radionuclide Therapy
  Other Names: PRRT
Drug: Capecitabine plus temozolamide — Chemotherapy
  Other Names: CAPE-TEM
  Arms: PRRT with Lu-177 DOTATATE PLUS Capecitabine-Temozolamide

SUMMARY:
Neuroendocrine tumours (NETs), better defined as neoplasms (NENs), are a heterogeneous group of neoplasms that range from well-differentiated tumours to more aggressive carcinomas. Peptide receptor radionuclide therapy (PRRT) with Lutetium-177 DOTATATE is the established standard of care for patients with well-differentiated metastatic or locally advanced GEP-NETs. It has demonstrated a significant improvement in outcomes compared to Octreotide LAR, both as a first-line and second-line treatment approach, following the results of NETTER-1 and NETTER-2 trials, respectively. ENETS guidelines recommend the use of Ga-68 labeled DOTANOC/TOC/TATAE imaging only for WHO Grade 1 NET whereas FDG PET is the preferred modality for WHO Grade 3 NEN and NEC. For Grade 2 tumors (Mib index ranging from 3-20%), there are no strong recommendations for the addition of FDG PETCT in existing diagnostic algorithm. FDG PET positivity has been shown to be an independent predictor of shorter progression-free and overall survival in NET patients undergoing peptide receptor radionuclide therapy (PRRT). (8) Consequently, it is imperative to address FDG-avid tumors by integrating PRRT and chemotherapy. There are no strong recommendations for the grade wise management of GEP-NETs particularly grade 2 & 3. Although recently published NETTER 2 trial substantiated the role of PRRT as a first line treatment for advanced grade GEP-NETs, still there is lack of evidence supporting the addition of chemotherapy in management of GEP-NETs. Given the absence of a prospective study to establish this treatment regimen, we designed a Phase 3 Randomized Controlled Trial to evaluate the combination of PRRT and CAPE-TEM-based chemotherapy in patients with FDG-positive metastatic well-differentiated NETs.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a heterogeneous group of malignancies ranging from well- differentiated, slowly growing tumors to poorly differentiated neoplasms, which are aggressive and less frequent. Neuroendocrine cells have the ability to express several peptide receptors in high volumes, especially somatostatin receptors, which are heptahelical G-protein-coupled glycoprotein transmembrane receptors. In the most recent SEER register (SEER-17), more than half of all NETs, i.e. 61%, were gastroenteropancreatic neuroendocrine tumors (GEP-NETs), with the highest frequency being found in the rectum (17.7%), the small intestine (17.3%), and the colon (10.1%) . The tumor biology varies with the location of the primary tumors as well as with the grade and staging of the tumors. The malignant potential ranges from the most benign types of tumor to small intestinal tumors and up to neuroendocrine carcinoma (NEC) with very malignant behavior. The tumors are graded according to the classification system of the World Health Organization (WHO), wherein a new classification system is just being accepted. The tumors are divided into grade 1 NET (NET-G1), with a proliferation <3%, NET-G2 with a proliferation between 3 and 20%, NET-G3, which is a new group with a Ki-67 >20%, and finally NEC-G3, exhibiting a Ki-67 of >20% as well (unpublished data). Of note, the difference between NET-G3 and NEC-G3 is mainly the degree of differentiation. NET-G3 are well-differentiated tumors, often with expression of somatostatin receptors. NEC-G3 are poorly differentiated tumors that usually lack expression of somatostatin receptors.

NETs are characterized by a general lack of symptoms until they are in advanced phase, and early biomarkers are not as available and useful as required. Heterogeneity is an intrinsic, pivotal feature of NETs that derives from diverse causes and ultimately shapes tumor fate. The different layers that conform NET heterogeneity include a wide range of distinct characteristics, from the mere location of the tumor to its clinical and functional features, and from its cellular properties, to the core signaling and (epi)genetic components defining the molecular signature of the tumor. The importance of this heterogeneity resides in that it translates into a high variability among tumors and, hence, patients, which hinders a more precise diagnosis and prognosis and more efficacious treatment of these diseases. Heterogeneity can be assessed objectively by molecular imaging techniques. Patients with well- differentiated GEP NETs undergo imaging with Ga-68-DOTATOC PET/CT (DOTA PET/CT), which is a somatostatin-receptor (SSTR)-specific imaging tracer. PET/CT with 68Ga-DOTA-peptides has been reported to present a higher sensitivity for the detection of well-differentiated, less aggressive NETs than well tolerated with negligible grade 3/4 toxicities. After a median follow-up period of 36 months, the median OS was not achieved with a median PFS of 48 months. At 3 months after completion of combination of PRRT and chemotherapy, 2% of patients showed a complete anatomical response, 28% a partial response, 68% stable disease, and only 2% progression. On FDG PET/CT, 27% achieved a complete metabolic response during the follow-up period. A biochemical response (>25% fall in chromogranin-A levels) was seen in 45%. These results established the effectiveness of the combination of PRRT and chemotherapy which is now practiced routinely. However, there is no prospective study to establish this treatment regime. The investigators therefore propose to prospectively evaluate the combination of PRRT and chemotherapy in patients with well-differentiated NETs, in a systematic manner to generate reliable conclusions with regards to this treatment regimen for intermediate to high grade NETs. On the other hand, 18F-FDG PET/CT is preferred for more aggressive, less differentiated NETs as there is emerging evidence that the presence of increased expression of GLUT (glucose-transporter) receptors in NETs highlights an increased propensity for invasion and metastasis, and an overall poorer prognosis. In fact, a strong association has recently been shown between higher 18F-FDG uptake and worse outcome even in patients with well-differentiated or low-grade tumors, with provision of prognostic information independently of the mitotic rate. Accordingly, 18F-FDG has an important role in managing patients with NETs because of its high prognostic value and its higher sensitivity in delineating disease extent, especially in aggressive and high-grade and aggressive intermediate-grade tumors. While DOTA PET avidity is a feature of well-differentiated disease, FDG avidity tends to be associated with more aggressive, de-differentiated disease. Grade 1 NET tends to be DOTA-avid but negative on FDG PET, whereas grade 3 NEC generally shows the opposite imaging phenotype. Grade 2 NET may demonstrate uptake of both tracers. Irrespective of pathological grade, the distribution of these tracers may not be spatially concordant, with some lesions having either DOTA or FDG avidity, but not both. This highlights the limitations of relying on histopathological grade from a single biopsy site to predict disease behavior. Despite the prognostic utility of pathological grading, FDG PET positivity has been consistently shown to be independently associated with a poor prognosis. SSTR expression on the surface of NET enables the use of somatostatin analogues labelled with particle-emitting radionuclides for targeted peptide receptor radionuclide therapy (PRRT) NETTER-1 trial has established Lu-177 PRRT as standard of care in treatment of metastatic well-differentiated GEP NETs. However, FDG positivity in these tumors suggests presence of aggressive phenotypes and warrants simultaneous use of chemotherapy. Strosberg et.al, have shown exceptionally high and durable response rate with combination of Capecitabine and temozolomide in metastatic well, or moderately differentiated pancreatic neuroendocrine tumor. Combination of PRRT and chemotherapy, that is, temozolomide-capecitabine (CAP-TEM) has been therefore effective in patients showing SSTR and GLUT receptor expression on Ga-68 DOTA PET and FDG PET respectively. Kong et al studied a retrospective cohort of 52 patients selected for treatment on the basis of somatostatin-receptor imaging without spatially discordant FDG-avid disease. All patients received conventional PRRT regimen, in addition oral capecitabine was added after every PRRT cycle. Clinical, biochemical and imaging response was assessed after completion of induction. Combination of PRRT and chemotherapy was well tolerated with negligible grade 3/4 toxicities. After a median follow-up period of 36 months, the median OS was not achieved with a median PFS of 48 months. At 3 months after completion of combination of PRRT and chemotherapy, 2% of patients showed a complete anatomical response, 28% a partial response, 68% stable disease, and only 2% progression. On FDG PET/CT, 27% achieved a complete metabolic response during the follow-up period. A biochemical response (>25% fall in chromogranin-A levels) was seen in 45%. These results established the effectiveness of combination of PRRT and chemotherapy which is now practiced routinely. However, there is no prospective study to establish this treatment regime. The investigators therefore propose to prospectively evaluate combination of PRRT and chemotherapy in patients with well-differentiated NETs, in systematic manner to generate reliable conclusion with regards to this treatment regimen for intermediate to high grade NETs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than 18 years
* Histopathological diagnosis of GEP-NET, necessarily satisfying all the the criteria below
* Well differentiated G2 (Ki67 : ≥3-20%) OR G3 (ki67- greater than 20-55%), OR
* Well-differentiated G1 (<3%) with disease progression in last 6 months
* Positive Ga-68-DOTANOC PET/CT, Krennings score >/=3
* Positive FDG PET imaging, grade 3 or 4 uptake
* Locally advanced/inoperable disease or metastatic disease
* Karnofsky performance-status score of at least 60 or ECOG performance status </= 2
* Life expectancy greater than 6 months

Exclusion Criteria:

* Serum creatinine level of more than 1.6 mg/dl or a creatinine clearance of less than 50 ml/min
* Hemoglobin level of less than 8.0 g per deciliter
* Red blood cell count noty less than 300,000/cubic millimeter White cell count of less than 2000 per cubic millimeter
* Platelet count of less than 75,000 per cubic millimetre
* Total bilirubin level of more than 3 times the upper limit of the normal range
* Serum albumin level < 3.0 g/dl
* Treatment with more than 30 mg of octreotide LAR within 4 weeks before randomisation.
* Peptide receptor radionuclide therapy at any time before randomisation
* Pregnancy and Lactation
* Patients with concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2027-08-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival (PFS) will be defined as the time from enrolment to the time of disease progression or death, or to the date of last tumor assessment (until 36 months from last day of completion of treatment) without any such event (censored observation).

SECONDARY OUTCOMES:
Overall survival | Time interval from enrolment to the date of death or last observation (censored), maximum until 24 months.
  The duration of overall survival (OS) will be determined by measuring the time interval from enrolment to the date of death or last observation (censored).
Quality of Life parameters | Day 1 of every treatment in both arms until treatment completion, and thereafter every 6 months upto 24 months
  QOL analysis will be conducted using the following tools (with appropriate language translations) EORTC QLQ-30 EORTC G.I.NET-21

CONTACTS AND LOCATIONS:
Overall Officials: Ameya Puranik, MD, Principal Investigator — Professor and Consultant
Locations (2):
- India (2):
  - Tata Memorial Hospital, Mumbai, India, Mumbai, Maharashtra
  - Advanced Centre for Treatment, Research and Education in Cancer (ACTREC), Navi Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parghane RV, Ostwal V, Ramaswamy A, Bhandare M, Chaudhari V, Talole S, Shrikhande SV, Basu S. Long-term outcome of "Sandwich" chemo-PRRT: a novel treatment strategy for metastatic neuroendocrine tumors with both FDG- and SSTR-avid aggressive disease. Eur J Nucl Med Mol Imaging. 2021 Mar;48(3):913-923. doi: 10.1007/s00259-020-05004-5. Epub 2020 Sep 2. PMID 32876706
- [Background] Nicolini S, Bodei L, Bongiovanni A, Sansovini M, Grassi I, Ibrahim T, Monti M, Caroli P, Sarnelli A, Diano D, Di Iorio V, Grana CM, Cittanti C, Pieri F, Severi S, Paganelli G. Combined use of 177Lu-DOTATATE and metronomic capecitabine (Lu-X) in FDG-positive gastro-entero-pancreatic neuroendocrine tumors. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3260-3267. doi: 10.1007/s00259-021-05236-z. Epub 2021 Feb 18. PMID 33604690
- [Derived] Puranik AD, Dev ID, Yadav S, Rangarajan V, Agrawal A, Basu S, Chaudhari VA, Ramaswamy A, Ostwal V, Bhandare MS, Shrikhande SV, Parghane RV, Bhargava P, Bal MM, Yadav S, Patkar S, Goel M, Purandare NC, Shah S, Choudhury S, Ghosh S, Venkatachalam M. PReCedeNT trial: Phase III randomized-controlled trial of Lutetium - 177 DOTATATE Peptide Receptor Radionuclide Therapy (PRRT) plus Chemotherapy versus PRRT alone in FDG-avid, Well-differentiated Gastroenteropancreatic neuroendocrine tumors (GEP-NETs). BMC Cancer. 2025 Oct 28;25(1):1659. doi: 10.1186/s12885-025-15111-x. PMID 41152774
- See also: Clinical Trial Registry of India — https://ctri.nic.in/Clinicaltrials/pubview.php

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT07185672/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT07185672/ICF_001.pdf